CLINICAL TRIAL: NCT06555939
Title: Promoting Resilience Among Adolescents and Young Adults With Sickle Cell Disease
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Children's Hospital (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Principal Investigator, Abby Rosenberg, Chief, Pediatric Palliative Care, Boston Children's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB-P00048890
Record Dates: First submitted 2024-08-13; First posted 2024-08-15 (Actual); Last update posted 2025-12-10 (Actual); Status verified 2025-12

CONDITIONS: Sickle Cell Disease
Keywords: adolescents; young adults; resilience; sickle cell disease; collaborative care
MeSH Terms: conditions — Anemia, Sickle Cell

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CoCM+PRISM (Experimental): Collaborative Care Model (CoCM) includes a care manager, a defined population of patents/registry for tracking inclusion and progress, validated patient-reported outcome measures, and weekly inter-professional team meetings. This arm includes the use of an inter professional team to triage, plan and deliver care. the PRISM intervention, a brief, skills-based program targeting 4 resilience resources, will be delivered 1:1 as part of this treatment arm.
  Interventions: Behavioral: Collaborative Care Model; Behavioral: Promoting Resilience in Stress Management

INTERVENTIONS:
Behavioral: Collaborative Care Model — The interprofessional team will meet weekly to review survey scores, endorsed psychological and physical health needs, as well as other concerns. They will conduct assessments as a group that may include referrals for additional support.
Behavioral: Promoting Resilience in Stress Management — PRISM targets 4 resilience resources: stress management, goal-setting, cognitive reframing and meaning-making. It is delivered one-on-one by trained coaches in English or Spanish via HIPAA compliant video-conference or in-person. Sessions are delivered every 1-2 weeks based on patient preference. To facilitate practice between sessions, all participants 13 or older have access to the digital PRISM app.
  Other Names: PRISM

SUMMARY:
Adolescents and young adults with sickle cell disease (SCD) face challenges managing their illness and maintaining their well-being. This study proposes to test the feasibility and acceptability of a resilience-promoting intervention through a Collaborative Care Model. The primary goal is to determine with the resilience intervention (PRISM) is feasible and acceptable for adolescents and young adults with SCD. Exploratory outcomes include whether this intervention improves depression, anxiety, and pain interference.

DETAILED DESCRIPTION:
Adolescents and Young Adults (AYAs) with blood disorders are at risk for poor physical, psychological, and social outcomes. Sickle Cell Disease (SCD) is a life-limiting condition, defined as a group of inherited red blood cell disorders disproportionally affecting non-Hispanic Black, African American, and Hispanic/Latino groups. AYAs with SCD experience racial bias, disease-related stigma, and under-treated symptoms, all of which translate to additional challenges managing their illness and maintaining their well-being. This study proposes to address the gaps of mental health support for youth with SCD through delivery of a resilience-promoting intervention (PRISM) using a Collaborative Care Model (CoCM). The primary objective of this study is to test the feasibility and acceptability of a collaborative care model to sustainably deliver the PRISM intervention for AYAs with SCD. Leveraging successful strategies implemented for patients with cancer, we will pilot-test this approach with N=25 AYAs in the Dana-Farber Cancer Institute/Boston Children's hospital (DFCI/BCH) SCD clinic. The primary outcome of interest is feasibility, defined as >50% enrollment. Secondary outcomes include patient reported outcomes of feasibility, acceptability, and satisfaction. Exploratory outcomes include assessment of depression, anxiety, and pain interference. We hypothesize this will be feasible and acceptable in this patient population.

ELIGIBILITY:
Inclusion Criteria:

* Aged ≥ 12 and ≤ 25 years of age at baseline
* Diagnosed with Sickle Cell Disease (HbSS, HbSC, HbS-Beta Thalassemia, and other related hemoglobinopathies)
* Receiving Medical Care at the DFCI/BCH Blood Disorders Center.
* Scored > 9 on Patient Health Questionnaire 9-item (PHQ-9) or Generalized Anxiety Disorder (GAD)
* Able to speak English or Spanish language (for PRISM sessions)
* Able to read English or Spanish language (for completion of surveys)
* Cognitively able to participate in PRISM sessions and complete written questionnaires and surveys, as judged by the site investigator
* Willing and able to adhere to the study visit schedule and other protocol requirements

Exclusion Criteria:

* does not meet above criteria

Ages: 12 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 25 (Estimated)
Dates: Start 2025-10-23 (Actual); Primary Completion 2029-09 (Estimated); Study Completion 2030-09 (Estimated)

PRIMARY OUTCOMES:
Enrollment rate (feasibility) | 3-months
  feasibility assessed by >50% enrollment rate

SECONDARY OUTCOMES:
Acceptability | 3-months post-enrollment
  program usefulness and willingness to recommend it (assessed via qualitative interviews)

OTHER OUTCOMES:
Patient-Health Questionnaire (PHQ-9) | 3-months
  depressive symptoms, range 0-27 with higher scores indicating higher symptoms
Generalized Anxiety Disorder (GAD-7) | 3-months
  anxiety symptoms, range 0-21 with higher scores indicating higher symptoms

CONTACTS AND LOCATIONS:
Locations (1):
- Boston Children's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
all deidentified IPD that underlie results in a publication
Supporting Information: Study Protocol, SAP
Time Frame: 6-months after manuscript is published
Access Criteria: contact PI